CLINICAL TRIAL: NCT05148975
Title: The Diagnosis of Superinfections in Mechanically Ventilated Covid-19 Patients
Acronym: SUPER-BAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Hudec, MD, physician, Brno University Hospital
Other Study IDs: 145/21
Record Dates: First submitted 2021-12-02; First posted 2021-12-08 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Pneumonia; Superinfection; ARDS, Human
Keywords: COVID-19; pneumonia; superinfection; bronchoalveolar lavage; ARDS
MeSH Terms: conditions — Superinfection; Respiratory Distress Syndrome; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Part of the sample from bronchoalveolar lavage fluid (BALF) will be frozen for possible further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild ARDS due to Covid- 19 pneumonia: Adults with SARS-CoV-2 PCR positivity in the last 21 days on mechanical ventilation for Covid-19 pneumonia, fulfilling criteria for mild acute respiratory distress syndrome (ARDS) definition.
  Interventions: Diagnostic Test: Bronchoalveolar lavage fluid diagnostics

INTERVENTIONS:
Diagnostic Test: Bronchoalveolar lavage fluid diagnostics — Bronchoalveolar lavage fluid diagnostics for superinfection in patients with COVID-19 pneumonia.

SUMMARY:
Patients with severe Coronavirus Disease 2019 (Covid-19) pneumonia depending on mechanical ventilation are at risk of superinfections, especially infections of respiratory tract. This multicententer prospective observational study is focused on early diagnosis of respiratory tract superinfections and identification of risk factors (immunosuppressive therapy,...). Investigators will use bronchoalveolar lavage fluid (BALF) for Polymerase Chain Reaction (PCR) detection of pathogens and antigenic detection of mycoses.

This project can support the routine use of BALF and PCR diagnostics for early detection of pathogens. Data will be compared with historical cohort of patients without routine BAL.

DETAILED DESCRIPTION:
Prospective, observational multicenter study

The inclusion criteria are as follows:

Age > 18 years Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) PCR positivity in the last 21 days Mechanical ventilation for Covid-19 pneumonia Presence of lung infiltrations on the chest X-ray or ground glass opacity, crazy paving or lung infiltrations on the chest CT Oxygenation disorder according to Acute Respiratory Distress Syndrome (ARDS) definition: Partial Pressure of Oxygen in Arterial Blood (PaO2) / fraction of inspired oxygen (FiO2) <300 mmHg with positive end expiratory pressure (PEEP) at least 5 cmH2O

The exclusion criteria are as follows:

Disagreement with the inclusion in the trial

Outcomes Primary outcome: incidence and characteristics of superinfections in patients with Covid-19.

Secondary outcome:

Markers of infection/inflammation diagnostic values for the diagnosis of a specific type of superinfection.

Comparison of the incidence of bacterial and opportunistic superinfections with a historical cohort, where the extension of diagnostics with bronchoalveolar lavage was performed only in patients who did not respond to antibacterial therapy

Size of the group of patients The number of patients enrolled in the study depends on the epidemiological situation and the number of admitted patients with severe Covid-19 disease. Investigators expect that the University Hospital at St. Anne's enrolls 75 patients and the University Hospital Brno also enrolls 75 patients. The size of the group is not relevant due to character of the study.

Monitored parameters Bronchoalveolar lavage (BAL) is the only procedure that differs from standard care. It is usually performed in patients with a suspected lung infection that does not respond to antibiotic therapy. In the study, BAL will be performed early after admission and then in 7-day intervals ( ± 1 day). This interval can be shortened to a minimum of 3 days if there are signs of a new lung infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* SARS-CoV-2 PCR positivity in the last 21 days
* Mechanical ventilation for Covid-19 pneumonia
* Presence of lung infiltrations on the chest X-ray or ground glass opacity, crazy paving or lung infiltrations on the chest CT
* Oxygenation disorder according to ARDS definition: PaO2 / FiO2 <300 mmHg with PEEP at least 5 cmH2O

Exclusion Criteria:

* Disagreement with the inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with COVID-19 ARDS on mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Superinfection incidence | 1 year
  The incidence and characteristics of superinfections in patients with Coronavirus Disease 2019 (COVID-19).

SECONDARY OUTCOMES:
The aasociation inflammation diagnostic values and the diagnosis of superinfection | 1 year
  Markers of infection / inflammation diagnostic values for the diagnosis of a specific type of superinfection.
The differention of superinfection diagnosis between historical cohort and actual cohort. | 1 year
  Comparison of the incidence of bacterial and opportunistic superinfections with a historical cohort, where the extension of diagnostics with bronchoalveolar lavage was performed only in patients who did not respond to antibacterial therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - University Hospital Brno, Brno, Czech Republic
  - St. Annes University Hospital, Brno, Czech Republic

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT05148975/Prot_000.pdf